CLINICAL TRIAL: NCT06148740
Title: An Investigation of the Effects of a Skin Serum Containing Propolis on Skin Health and Appearance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manuka Health (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20376
Record Dates: First submitted 2023-11-19; First posted 2023-11-28 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Skin Health
MeSH Terms: interventions — Propolis; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pro Vitality Daily Restorative Face Serum (Experimental): Participants will be required to apply the test product in the morning and before sleeping at night.
  After thoroughly cleansing and toning the face, the participants will apply 2-3 drops onto clean dry fingers and massage over the entire face until fully absorbed.
  The product should be followed with the participants' preferred moisturizer.
  Interventions: Other: Manuka Health Pro Vitality Daily Restorative Face Serum with Propolis & Vitamin C

INTERVENTIONS:
Other: Manuka Health Pro Vitality Daily Restorative Face Serum with Propolis & Vitamin C — Skin serum containing propolis, vitamin C, and manuka honey.

SUMMARY:
This is a virtual, single-group clinical trial that will last 8 weeks. Participants will use the Manuka Health Pro Vitality Daily Restorative Face Serum with Propolis & Vitamin C twice daily and complete questionnaires at Baseline, Week 2, Week 4, and Week 8. Participants will also undergo skin analysis via the Optic Elite facial skin analysis system at Baseline and Week 8.

ELIGIBILITY:
Inclusion Criteria:

* Female between 30-42 years of age.
* Must be in good general health.
* Must have concerns with overall skin health and appearance, including:

Spots or blemishes Uneven skin tone Dull-looking skin

* Must be using the same cleanser, toner, and moisturizer for at least one month prior to starting the study.
* Must be willing to keep using the same cleanser, toner, and moisturizer for the duration of the study.
* Must not be using oral or topical retinoids.
* In the last three months, has not introduced any new medications or supplements that target skin health.
* Must be willing to comply with the protocol.

Exclusion Criteria:

* Anyone with an allergy to bees or bee products.
* Females who are pregnant or breastfeeding.
* Unwilling to follow the protocol.
* Unwilling to maintain use of the same cleaner, toner, and moisturizer for the duration of the study.
* Currently participating in another study.
* Use of oral or topical retinoids.
* Individuals with cystic acne or otherwise self-reported very acne-prone skin.
* Use of a prescription medication relevant to the skin.
* Anyone undergoing cosmetic procedures during the study, including Botox, laser, or chemical peel treatments.
* Anyone sensitive or allergic to any ingredients found in the products.
* Anyone with severe chronic conditions, including oncological conditions, psychiatric disorders or diabetes.

Ages: 30 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-11-09 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Changes in signs of skin health over time assessed via Optic Elite Skin Analysis. [Timeframe: Baseline to Week 8] | 8 weeks
  The Optic Elite skin analysis system clinically measures the surface and subsurface layers of skin using digital imaging technology. Participants will receive a score that can be compared between time points.

SECONDARY OUTCOMES:
Changes in self-perceived skin clarity. [Timeframe: Baseline to Week 8] | 8 weeks
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.
Changes in self-perceived skin hydration. [Timeframe: Baseline to Week 8] | 8 weeks
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.
Changes in self-perceived skin texture. [Timeframe: Baseline to Week 8] | 8 weeks
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.
Changes in self-perceived skin pigmentation. [Timeframe: Baseline to Week 8] | 8 weeks
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.
Changes in self-perceived skin irritation. [Timeframe: Baseline to Week 8] | 8 weeks
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.
Changes in self-perceived skin brightness.[Timeframe: Baseline to Week 8] | 8 weeks
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.
Changes in self-perceived skin tone evenness. [Timeframe: Baseline to Week 8] | 8 weeks
  Measured via study-specific questionnaires using a 5-point Likert scale. A lower score indicates a more favourable response, with 0=Not noticeable and 4=Severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided